CLINICAL TRIAL: NCT02443038
Title: Yoga's Effect on Fall Risk Factors in the Rural, Older Adult Population; an Academic/Community Partnership
Acronym: Yoga/Falls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WPP2774
Record Dates: First submitted 2015-04-17; First posted 2015-05-13 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Patient Fall
Keywords: patient fall; yoga; balance
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home Exercise (Active Comparator): Participants will practice 10 minutes of yoga in addition to 5 minutes of relaxation exercises at home each day when not in class.
  Interventions: Other: Yoga
- Relaxation Exercise (Placebo Comparator): Participants will practice 5 minutes of relaxation exercises at home each day when not in class.
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — 16 bi-weekly 50-60 minute yoga classes, followed by daily, 10 minute home exercise poses and 5 minute relaxation, the control group will practice 5 minutes relaxation, each day between classes.
  The first of 3 classes is the 8-10 member advisory board, the second and third classes with 10-15 participants in each workshop will be held in other counties. There will be 2-3 months between the first set of classes and second and third set of classes to refine methods and conduct enrollment and testing for the subsequent groups.

SUMMARY:
This is a 2 year pilot/feasibility project to develop an intervention, test research methods, and evaluate the effects of yoga on core strength and balance of an older rural population in an effort to ultimately reduce the frequency of falls. The investigators' goal for this project is for community and academic partners to develop a yoga program that is feasible, safe, and acceptable to an older adult population, then test the program, research methods and evaluation, in preparation for conducting a larger randomized trial of the intervention.

DETAILED DESCRIPTION:
This is a 2 year pilot project to develop an intervention, and to test research methods and evaluation to assess the effects of yoga on core strength and balance of an older population in an effort to ultimately reduce the frequency of falls. The literature suggests that increased core body strength improves balance and reduces fall frequency in the elderly. Yoga increases core strength. There is limited evidence that regular yoga exercising is associated with a decreased frequency of falls in the older adult population. However, there have not been any randomized trials testing the impact of a yoga program on fall frequency. The investigators' goal for this project is to develop a yoga program that is feasible, safe, and acceptable to an older population then test the intervention, research methods and evaluation in preparation for conducting a randomized trial of the intervention.

This study is conducted with the investigators community partner, the aging and disabilities resource center (ADRC) of Southwest Wisconsin. The ADRC will help with recruiting, posting on ADRC's website and flyers. The ADRC will provide locations for classes and assessments. Recruitment will also occur through local community event announcements.

An advisory board of 8-10 members of older adults will inform about needs and feasibility, and help review the handbook and video. The advisory boards involvement will be in the preparatory phase of the research, along with full project oversight.

Enrollment Questionnaire

Eligible subjects will be asked to complete a brief questionnaire. The questionnaire will include questions about: 1) Demographics including age, gender, race, ethnicity, years of education, income level, 2) Number of falls in the past 1 month, 6 months and 1 year, and 3) Fear of falling questions using the ABC (Activities-specific Balance Confidence Scale).

Visit 2- Physical Activity Assessment

The physical activity assessment will be conducted one-on-one by a Physical Therapist and occur at the individual ADRC offices where yoga classes will be held. Height and weight will be measured during the first assessment only. Testing will consist of 3 low physical demand tests of static and dynamic balance and gait characteristics: 1) The Berg Balance Scale, 2) The Functional Gait Assessment, and 3) The Dynamic Gait Index. Each of these tests requires a minimal to moderate amount of exertion, typically not enough to cause any shortness of breath with transient mild increase in heart rate. The total time anticipated to conduct the testing is 60 minutes.

The investigators chose these tests because they are validated measures for the investigators' subject population, do not require any special equipment, take only a few minutes to administer, and are safe to perform in an older adult population.

Visits 3 to 18- Intervention

The intervention consists of 16 bi-weekly 50-60 minute yoga classes, conducted by certified yoga therapists, and in case of the advisory group, after classes questions about improvement of classes that will take about 5 minutes. Additionally, 10 minute home exercise poses and 5 minute relaxation will be done each day between classes. The control group will practice 5 minutes relaxation on days between classes.

There will be 3 classes (in 3 different counties), the first is the 8-10 member advisory board. The second and third classes will have 10-15 participants in each workshop. The target is up to 60 total participants (including advisory board). There will be 2-3 months between the first set of classes and second and third set of classes to refine methods and conduct enrollment and testing for the subsequent groups.

A co-investigator will give out envelopes that contain the patient assignment to home practice or no home practice during the 3rd visit. The envelopes will be numbered and participants will randomly choose among the envelopes. The co-investigator will note the participant name and the envelope number but will not know the content of the envelope with the assignment. Another investigator will have noted the assignment to home exercise or control and the envelope number in a file that will be saved on a password protected computer in the investigators office and backed up on a UW- Madison secured server. A printout will be placed in a sealed envelope and kept in a locked ADRC office to be opened upon completion of data collection.

The general philosophy of the yoga classes is to create an environment of safety during all poses and avoid a culture of competition or subjects pushing themselves beyond individual abilities. Classes will consist of: 1) Centering; 2) Warm up; 3) A variety of simple poses with modifications to increase safety and reduce potential for falls (pictures of examples included in the manual as described/illustrated below, including 3 home practice poses; 4) cool down; and 5) 5 minute relaxation period. Poses will focus on alignment principles, lower extremity and core strengthening, and common flexibility deficits thought to be related to impaired balance. Modifications for individual range of motion will be provided as necessary. Poses will be supplemented or advanced to accommodate individual needs.

Subjects (intervention group) will also be asked to perform a set of poses at home taking approximately 10 minutes each day. The poses will be illustrated with photos in the home log. The home exercises will be performed daily each week on days other than class days. Subjects will record home activity as below.

Home Log Book and Data Collection, during the Intervention

Subjects (intervention group) will be given a home log book at the first yoga class. The log book includes general instructions, researcher contact information and specific instructions for the 3 home poses including picture illustrations. Subjects will be instructed to record the date and length of time each time the subjects do home poses and any discomfort or problems that occur with home exercises. Poses will be supplemented or advanced to accommodate individual needs. Subjects will be instructed to bring the log books to each class so instructors can check to see if the log books are being completed correctly and assess for any adverse events (AEs) and unanticipated problems (UPs).

Subjects will also track falls during the 8 week intervention and the 4 months following the completion of the intervention.

Home Log study control group

Half of the class will be randomized into either a home exercise group or a control group which will not do any yoga exercises outside of the classroom environment. The control group will be encouraged to do the yoga poses learned in class at home after the class is complete.

Instructors will record subject attendance at each class, if the subjects brought log book and AEs or UPS. Instructors will also record total class time from start to finish and all the poses done during the class into a spreadsheet.

The investigators anticipate that total twice weekly yoga classes will take 16 hours and the home activities will take about (5 x 15 minutes x 16 weeks) 20 total hours for the group assigned to home exercises and (5 x 5 minutes x 16 weeks) about 6.5 hours for the control group. Total time involvement including 16 hours of class time, enrollment visit and pre and post assessment visits is about 40 hours for the intervention group and 26 hours for the control group.

Visit 19- Repeat Physical Assessment and Questionnaire

Final assessment will occur within 2 weeks of the final yoga class. Instructors and investigators will strongly encourage all participants, including drop outs, to complete the final assessment. Final assessment will include: 1) A questionnaire with the pre-intervention falls related survey questions (including the ABC (Activities-specific Balance Confidence Scale), additional questions about the yoga classes, home exercises and use of the logbook; 2) Post-intervention physical activity assessment. The post-intervention physical assessment is the same as the initial assessment except the height and weight are not re-measured. This final visit is expected to last about 1 hour.

A co-investigator will call participants 2 months and 4 months after completing the class, to ask questions about falls and yoga practice at home. Each phone call will take about 5 minutes.

Sample Size and Analysis:

Since this is a pilot program to develop the intervention and assessment methods, the investigators sample size of up to 60 subjects is based on practicality and limited by available time and funding. Based on previous yoga teaching experience, 14 people is a manageable class size to allow for personal attention to adjust poses as necessary for subject safety for each of the groups. The investigators anticipate 20% drop out rate with a final sample size of up to 48 subjects. With this small sample size, and moderate level of pre-intervention physical function of the subjects, the investigators may not find significant changes in the physical activity measures. The investigators do hope to find some trend toward increased ability to maintain balance. Descriptive statistics will be used to create summed scores for fall questions. Paired tests and repeated-measures analysis of variance (ANOVA) will be used to analyze the pre- intervention and post- intervention physical activity measures.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. Age 60 and older
3. Able to walk 150 feet without assistive devices such as a cane or walker. This is a commonly used definition of an "independent ambulator" according to the Functional Independence Measure.
4. Cognitively intact as evidenced by correct answers to the mini-cogMemory Impairment Screen.
5. Able to provide informed consent.

Exclusion Criteria:

1. Pelvic or lower extremity injury in the previous 6 months that required temporary use of an assistive device, including crutches, for more than 7 days.
2. Pelvic or lower extremity orthopedic surgery in the previous 12 months.
3. Cardiac or other medical condition with previous physician instructions to avoid low intensity exercise.
4. Neurologic condition that impairs strength or balance including herniated lumbar disc with nerve root compression, previous stroke with residual lower extremity weakness, Parkinson's Disease, Multiple Sclerosis, muscular dystrophy and other neuromuscular diseases.
5. Terminal condition with rapid progression of disease and not expected to live 6 months or more.
6. Inability to provide informed consent
7. Practiced yoga at home or in a classroom setting in the past 6 months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
occurence of falls | 6 months
  incidence and number of falls that occur for participants during the study

SECONDARY OUTCOMES:
Improved Balance | 6 months
  validated balance testing including the Berg Balance Scale, and testing of walking performance using the Functional Gait Assessment at the beginning and end of program.
qualitative information about feasibility of yoga in rural older adults | 6 months
  survey and discussion with participants and advisory board members
time to first fall | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Irene Hamrick, MD, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - Aging and Disability Resource Center- Iowa and Lafayette Counties, Dodgeville, Wisconsin
  - Aging and Disability Resource Center-Green County, Monroe, Wisconsin
  - Aging and Disability Resource Center-Grant County, Platteville, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
We plan to share our data after analysis and peer review of publication

REFERENCES:
- [Background] Berg K, Wood-Dauphinee S, Williams JI. The Balance Scale: reliability assessment with elderly residents and patients with an acute stroke. Scand J Rehabil Med. 1995 Mar;27(1):27-36. PMID 7792547
- [Background] Brown KD, Koziol JA, Lotz M. A yoga-based exercise program to reduce the risk of falls in seniors: a pilot and feasibility study. J Altern Complement Med. 2008 Jun;14(5):454-7. doi: 10.1089/acm.2007.0797. No abstract available. PMID 18564950
- [Background] Chiu YP, Fritz SL, Light KE, Velozo CA. Use of item response analysis to investigate measurement properties and clinical validity of data for the dynamic gait index. Phys Ther. 2006 Jun;86(6):778-87. PMID 16737403
- [Background] CDC. (2009). http://www.cdc.gov/injury/wisqars/fatal_injury_reports.html
- [Background] DiBenedetto M, Innes KE, Taylor AG, Rodeheaver PF, Boxer JA, Wright HJ, Kerrigan DC. Effect of a gentle Iyengar yoga program on gait in the elderly: an exploratory study. Arch Phys Med Rehabil. 2005 Sep;86(9):1830-7. doi: 10.1016/j.apmr.2005.03.011. PMID 16181950
- [Background] Gillespie LD, Robertson MC, Gillespie WJ, Sherrington C, Gates S, Clemson LM, Lamb SE. Interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD007146. doi: 10.1002/14651858.CD007146.pub3. PMID 22972103
- [Background] Hausdorff JM, Rios DA, Edelberg HK. Gait variability and fall risk in community-living older adults: a 1-year prospective study. Arch Phys Med Rehabil. 2001 Aug;82(8):1050-6. doi: 10.1053/apmr.2001.24893. PMID 11494184
- [Background] Hornbrook MC, Stevens VJ, Wingfield DJ, Hollis JF, Greenlick MR, Ory MG. Preventing falls among community-dwelling older persons: results from a randomized trial. Gerontologist. 1994 Feb;34(1):16-23. doi: 10.1093/geront/34.1.16. PMID 8150304
- [Background] Keith RA, Granger CV, Hamilton BB, Sherwin FS. The functional independence measure: a new tool for rehabilitation. Adv Clin Rehabil. 1987;1:6-18. No abstract available. PMID 3503663
- [Background] Kerrigan DC, Lee LW, Collins JJ, Riley PO, Lipsitz LA. Reduced hip extension during walking: healthy elderly and fallers versus young adults. Arch Phys Med Rehabil. 2001 Jan;82(1):26-30. doi: 10.1053/apmr.2001.18584. PMID 11239282
- [Background] Kerrigan DC, Todd MK, Della Croce U, Lipsitz LA, Collins JJ. Biomechanical gait alterations independent of speed in the healthy elderly: evidence for specific limiting impairments. Arch Phys Med Rehabil. 1998 Mar;79(3):317-22. doi: 10.1016/s0003-9993(98)90013-2. PMID 9523785
- [Background] Krishnamurthy M, Telles S. Effects of Yoga and an Ayurveda preparation on gait, balance and mobility in older persons. Med Sci Monit. 2007 Dec;13(12):LE19-20. No abstract available. PMID 18049442
- [Background] Lipton RB, Katz MJ, Kuslansky G, Sliwinski MJ, Stewart WF, Verghese J, Crystal HA, Buschke H. Screening for dementia by telephone using the memory impairment screen. J Am Geriatr Soc. 2003 Oct;51(10):1382-90. doi: 10.1046/j.1532-5415.2003.51455.x. PMID 14511157
- [Background] Oken BS, Zajdel D, Kishiyama S, Flegal K, Dehen C, Haas M, Kraemer DF, Lawrence J, Leyva J. Randomized, controlled, six-month trial of yoga in healthy seniors: effects on cognition and quality of life. Altern Ther Health Med. 2006 Jan-Feb;12(1):40-7. PMID 16454146
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Ross A, Thomas S. The health benefits of yoga and exercise: a review of comparison studies. J Altern Complement Med. 2010 Jan;16(1):3-12. doi: 10.1089/acm.2009.0044. PMID 20105062
- [Background] VanSwearingen JM, Paschal KA, Bonino P, Yang JF. The modified Gait Abnormality Rating Scale for recognizing the risk of recurrent falls in community-dwelling elderly adults. Phys Ther. 1996 Sep;76(9):994-1002. doi: 10.1093/ptj/76.9.994. PMID 8790277
- [Background] Wolfson L, Whipple R, Amerman P, Tobin JN. Gait assessment in the elderly: a gait abnormality rating scale and its relation to falls. J Gerontol. 1990 Jan;45(1):M12-9. doi: 10.1093/geronj/45.1.m12. PMID 2295773
- [Background] Wrisley DM, Kumar NA. Functional gait assessment: concurrent, discriminative, and predictive validity in community-dwelling older adults. Phys Ther. 2010 May;90(5):761-73. doi: 10.2522/ptj.20090069. Epub 2010 Apr 1. PMID 20360052
- [Background] Wrisley DM, Marchetti GF, Kuharsky DK, Whitney SL. Reliability, internal consistency, and validity of data obtained with the functional gait assessment. Phys Ther. 2004 Oct;84(10):906-18. PMID 15449976